CLINICAL TRIAL: NCT03876327
Title: Fecal Microbiota Transplantation As a Potential Treatment for Parkinson's Disease: A Pilot Study
Brief Title: Fecal Microbiota Transplantation As a Potential Treatment for Parkinson's Disease
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Soroka University Medical Center (Other)
Responsible Party: Principal Investigator, ARIK SEGAL MD, Principal Investigator, Soroka University Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0266-15-SOR
Record Dates: First submitted 2019-02-20; First posted 2019-03-15 (Actual); Last update posted 2020-08-05 (Actual); Status verified 2020-08

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: 3 groups were included in the study:
  1. PD patients that will undergo FMT tretment and a half of year follow-up-15 patients.
  2. PD patients that will not undergo FMT procedure and will donate stool sample only once-35 patients.
  3. healthy PD relatives, that live with them and have similiar life styling and which will donate stool sample only once-50 participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PD patients that will receive FMT (Experimental): fecal microbial transplantation once at the beginning of the study-15 patients.
  Interventions: Procedure: fecal microbial transplantation
- PD patients that will not receive FMT (No Intervention): do not receive treatment-35 patients.
- healthy people live with PD patients (No Intervention): do not receive treatment-50 participants.

INTERVENTIONS:
Procedure: fecal microbial transplantation — Fecal microbiota transplantation (FMT) is a technique in which intestinal microbiota are transferred from a healthy donor to the patient, with as primary goal to introduce - or restore - a stable and 'healthy' microbial community in the gut.
  Arms: PD patients that will receive FMT

SUMMARY:
this pilot study aims to further explore the potential usage of Fecal microbiota transplantation in treating constipation and possibly also motor symptoms in Parkinson's disease (PD) patients, and to increase understanding of the potential relationship between the identities of intestinal microbial communities and PD.

DETAILED DESCRIPTION:
Fecal microbiota transplantation (FMT) is a technique in which intestinal microbiota are transferred from a healthy donor to the patient, with as primary goal to introduce - or restore - a stable and 'healthy' microbial community in the gut.

Parkinson's disease (PD) is a neurodegenerative disorder characterized by motor symptoms and Gastrointestinal dysfunction, in particular constipation, affects up to 80% of PD patients and may precede the onset of motor symptoms by years.

this study include one group of PD patients that will receive FMT. two other groups will serve as controls:

1. PD patients that will not receive FMT
2. healthy people who live with PD patients in the same house and share similar surrounding

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged > 50 years, diagnosed as suffering from PD and under follow up of the Movement Disorders Clinic in Soroka University Medical Center.
* Subjects complaining of constipation .
* Subjects who did not perform a screening colonoscopy for colon cancer.
* Subjects who are clinically undertreated according to last Movement Disorders specialist's impression at the clinic visit.

Exclusion Criteria:

* Subjects who do not complain of constipation or seem clinically stable properly treated pharmacologically.
* Subjects who already underwent a screening colonoscopy for colon cancer.
* Subjects who suffer from a cognitive decline and could not give their consent, or patients who refuse to undergo a colonoscopy.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-08-19 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
motor parkinsonian symptoms | Change from baseline motor difficulties at 6 months
  motor symptoms assessed by UPDRS III questionaire
constipation level | Change from baseline constipation level at 6 months
  constipation will be assessed by a scoring system questionaire. 6 parameters are reviewed as scored fro 0 (mild symptom) to 4 (srvere symptom).

CONTACTS AND LOCATIONS:
Overall Officials: arik segal, MD, Principal Investigator — SOROKA MC
Locations (1):
- Soroka Medical Center, Beersheba, Israel

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Segal A, Zlotnik Y, Moyal-Atias K, Abuhasira R, Ifergane G. Fecal microbiota transplant as a potential treatment for Parkinson's disease - A case series. Clin Neurol Neurosurg. 2021 Aug;207:106791. doi: 10.1016/j.clineuro.2021.106791. Epub 2021 Jun 30. PMID 34237681